CLINICAL TRIAL: NCT01300780
Title: Effect of Preoperative Use of an Anti-inflammatory on Tooth Sensitivity Caused by In-office Bleaching: A Randomized, Double-blind Clinical Trial
Brief Title: Effect of an Anti-inflammatory on Tooth Sensitivity Caused by Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eloisa Andrade de Paula (Other)
Collaborators: Universidade Estadual de Ponta Grossa (Other); Fundação Araucária (Other)
Responsible Party: Sponsor-Investigator, Eloisa Andrade de Paula, Doctor, Universidade Estadual de Ponta Grossa
Organization: Universidade Estadual de Ponta Grossa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17838/2010
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Color Changes During Tooth Formation
Keywords: bleaching agent; tooth bleaching; sensibility
MeSH Terms: interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Active Comparator): The participants from the placebo group received a placebo (Talco pharma SM-200-Henrifarma produtos químicos e farmacêuticos LTDA, São Paulo, SP, Brazil) and participants from the etoricoxib group received a dose of a selective COX- 2 inhibitor etoricoxib 60 mg (Arcoxia, MSD, Campinas, SP, Brazil). All the participants were watched to ensure that they took the drugs or placebo 1 h before treatment. The drugs were similar in appearance. A second dose of placebo or etoricoxib (60 mg) was administered 24 h after the first dose. At the time the participants were required to take the second dose of the medicine, the research auxiliary called him/her and asked him/her to take the medicine.
  Interventions: Drug: Etoricoxib
- placebo group (Placebo Comparator): The participants from the placebo group received a placebo (Talco pharma SM-200-Henrifarma produtos químicos e farmacêuticos LTDA, São Paulo, SP, Brazil) and participants from the etoricoxib group received a dose of a selective COX- 2 inhibitor etoricoxib 60 mg (Arcoxia, MSD, Campinas, SP, Brazil). All the participants were watched to ensure that they took the drugs or placebo 1 h before treatment. The drugs were similar in appearance. A second dose of placebo or etoricoxib (60 mg) was administered 24 h after the first dose. At the time the participants were required to take the second dose of the medicine, the research auxiliary called him/her and asked him/her to take the medicine.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Etoricoxib — Group 2 - experimental Etoricoxib will receive two doses of selective anti-inflammatory to enzyme cyclooxygenase 2 (COX-2) (Etoricoxib 60 mg) given once every 24 hours;
  Other Names: Anti-inflamatory
  Arms: Experimental
Other: Placebo — Group 1 - Control Group will receive two doses of placebo tablet administered a every 8 hours,
  Other Names: Placebo group
  Arms: placebo group

SUMMARY:
Perhaps the use of a more selective anti-inflammatory drug, capable of inhibiting enzyme specific for pain may be more effective in preventing the tooth sensitivity caused by the inflammatory response produced by in-office bleaching. To the extent of the authors´ knowledge, no study has so far addressed the use of a selective anti-inflammatory drug specific for pain enzyme on tooth sensitivity, being this the aim of the present investigation.

DETAILED DESCRIPTION:
Study design This was a randomized, triple-blind, placebo-controlled, parallel-group clinical trial, with an equal allocation rate to receive either one of two treatments. The study took place in the clinic of the Brazilian Association of Dentistry in Guarapuava, Paraná from August 2010 to December 2010.

Inclusion and exclusion criteria

Patients included in this clinical trial were at least 18 years old and had good general and oral health. Participants were recruited by means of radio and TV advertisement. A total of 247 participants were examined in a dental chair to check whether they met the inclusion and exclusion criteria. The participants were required to have six caries-free maxillary anterior teeth, without resto- rations on the labial surfaces. The central incisors had to be shade C2 or darker as judged by comparison with a value- oriented shade guide (Vita Lumin, Vita Zahnfabrik, Bad Säckingen, Germany). Participants who had undergone tooth-whitening procedures, presented anterior restorations, were pregnant/lactating, had severe internal tooth discoloration (tetracycline stains, fluorosis, and pulpless teeth), were taking any type of medicine, had bruxism habits, or any other pathology that could cause sensitivity (such as recession and dentin exposure) were excluded from the study, since they would not be immediately eligible for a cosmetic treatment, such as bleaching. Participants who reported some earlier or present health problems in the stomach, heart, kidney and liver, or participants continuously using any with anti-inflammatory and antioxidant action were excluded from the study. Sample size calculation The primary outcome of this study was the absolute risk of TS. The absolute risk of TS was reported to be approximately 86 % for the bleaching product Whiteness HP Maxx (FGM, Joinville, SC, Brazil). Thus, 30 patients were required to have an 80 % chance of detecting, as significant at the two-sided 5 % level, a de- crease in the primary outcome measure from 86 % in the control group to 41 % in the experimental group.

Study intervention

Participants were randomly stratified by sex into the placebo and etoricoxib groups. The randomization process was performed by computer-generated tables by a third person not involved in the research protocol. Details of the allocated groups were recorded on cards contained in sequentially numbered, opaque, sealed envelopes. These were prepared by a third person not involved in any of the phases of the clinical trial. Once the participant was eligible for the procedure, and completed all baseline assessments, the allocation assignment was revealed by this envelope being opened by the mentioned third person. Neither the participant nor the operator knew the group allocation, both being blinded to the protocol.

The participants from the placebo group received a placebo (Talco pharma SM-200-Henrifarma produtos químicos e farmacêuticos LTDA, São Paulo, SP, Brazil) and participants from the etoricoxib group received a dose of a selective COX- 2 inhibitor etoricoxib 60 mg (Arcoxia, MSD, Campinas, SP, Brazil). All the participants were watched to ensure that they took the drugs or placebo 1 h before treatment. The drugs were similar in appearance. A second dose of placebo or etoricoxib (60 mg) was administered 24 h after the first dose. At the time the participants were required to take the second dose of the medicine, the research auxiliary called him/her and asked him/her to take the medicine. This procedure was implemented to increase adherence to the protocol.

The gingival tissue of the teeth to be bleached was isolated using a light-polymerized resin dam (Top Dam, FGM, Joinville, SC, Brazil). The 35 % hydrogen peroxide gel (Whiteness HP Maxx, FGM) was used in three 15-min applications for both groups in accordance with the manufacturer's directions. The in-office bleaching agent was refreshed every 15 min during the 45-min application period. Two bleaching sessions with 1 week interval between them were performed. All participants were instructed to brush their teeth regularly using fluoridated toothpaste (Sorriso Fresh, Colgate- Palmolive, São Paulo, SP, Brazil).

Shade evaluation

Shade evaluation was recorded before and 30 days after the bleaching treatment using two methods: subjective evaluation using a shade guide (Vita Lumin, Vita Zahnfabrik, Bad Säckingen, Germany) and an objective evaluation using the spectrophotometer (Easyshade, Vident, Brea, CA).

For the subjective examination, the 16 shade guide tabs were arranged from highest (B1) to lowest (C4) value, so that the color C2 was set. Although this scale is not linear in the truest sense, the changes were treated as though they represented a continuous and approximately linear ranking for the purpose of analysis. The measurement area of interest for shade matching was the middle one third of the facial surface of the anterior central incisor. For calibration purposes, five patients who were not included in the sample because they were used in the pilot study, participated in the training phase of this study. The two examiners, blinded to the allocation assignment, scheduled these patients for bleaching and evaluated their teeth against the shade guide at baseline and 30 days after the procedure. The two examiners were required to have an agreement of at least 85 % (Kappa statistic) before beginning the study evaluation. For the objective evaluation, a preliminary impression of the maxillary arch was made using dense silicone Adsil (Vigodent S/A Indústria e Comércio, Rio de Janeiro, RJ, Brazil). The impression was extended to the maxillary canine and served as a standard color measurement guide for the spectrophotometer. A window was created on the labial surface of the molded silicone guide for the central incisor to be evaluated. The window was made using a metal device with well-formed borders, with a radius of 3 mm. Only one operator took all the measurements in all 30 patients, using Vita Easyshade (Easyshade, Vident, Brea, CA) before and 30 days after the bleaching therapy. The shade was determined using the parameters of the Easyshade device where the following values were indicated: L*, (a*), and (b*), in which L* represents the value from 0 (black) to 100 (white) and a* and b* represent the shade, where a* is the measurement along the red-green axis and b* is the measurement along the yellow-blue axis. The color comparison before and after treatment is given by the difference between the two colors (ΔE), which is calculated using the formula: ΔE=((ΔL*)2+(Δa*)2+(Δb*) 2)1/2.

TS evaluation

The patients recorded their perception of TS during the first and second bleaching sessions using three pain scales. A 5-point verbal rating scale (0 = none, 1 = mild, 2 = moderate, 3 = considerable, and 4 = severe], a 0 to 100 numerical rating scale and a visual analogue scale using a 10-cm horizontal line with words "no pain" at one end and "worst pain" at the opposite end were used in this study. Subjects were asked to record whether they experienced TS during the treatment up to 1 h after, from 1 to 24 h and from 24 to 48 h after bleaching. The worst scores/numerical values obtained in both bleaching sessions were considered for statistical purposes. The values were arranged into two categories: percentage of patients that reported TS at least once during treatment (absolute risk of TS) and overall TS intensity.

Statistical analysis

The analysis was performed after the intention-to-treat protocol and involved all participants who were randomly assigned. The statistician was blinded to the study groups. The agreement between the examiners' objective evaluation was evaluated using the kappa statistic. The primary outcome absolute risk of TS was compared by using the Fisher's exact test at a 5 % level of significance. The relative risk as well as the confidence interval for the effect size was calculated.

TS intensity (secondary outcome) was also statistical- ly analyzed. The mean/median and standard deviation/interquartile range of the three pain scales were calculated. Color change, another secondary endpoint, was used to assess the efficacy of the bleaching treatment. For subjective evaluation, the means and standard deviations of SGU at baseline and 30 days after bleaching for each group were calculated. In order to evaluate whether the bleaching therapies were effective or not, the data from SGU of both groups were submitted to a two-way repeated measures ANOVA. A post-hoc analysis (Tukey's test) was used to make pairwise comparisons. The ΔL, Δa, Δb, and ΔE values were evaluated by Student's t test.

The data sets were plotted on histograms and inspected for normal distributions. Some data did not appear to be normally distributed, and therefore, nonparametric statistical tests were used to compare the various treatments. Statistical analyses of three pain scales comparing the two groups at the three different assessment points were performed using the Mann- Whitney U test. Comparisons between times within each group were performed using the Friedman tests. In all statistical tests, the significance level was set at p = 0.05 values less than or equal to 5 % indicated significant differences.

ELIGIBILITY:
Inclusion Criteria:

* will be included patients 18 years old and over
* with good general and oral health
* with the eight upper front teeth free of cavities and restorations in the buccal cavity

The initial color of those teeth must be C2 or dark, comparing with scale Vita Lumin (Vita Zahnfabrik, Bad Säckingen, Germany) organized in order of value.

Exclusion Criteria:

* shall be excluded patients who underwent any previous form of bleaching procedure
* lactating and pregnant patients
* who relates sensitivity
* severe dental browning (tetracycline staining, fluorosis or endodontics)
* with parafunctional habit or any other type of oral disease

Still will be excluded patients who have systemic conditions as stomach problems, heart, kidney and liver, or using any continuous drug with anti-inflammatory and antioxidant action.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Sensibility | Evaluation of sensibility during the tooth whitening and 24/48 after of the bleaching
  The effect of the product will be evaluated immediately, 1 Hour, 24 and 48 hours after the teeth bleaching applied to the patients, using a verbal scale of 5 points, also a numerical scale of 101 points will be used, In addition to these two scales a Visual Analogue Scale (VAS, which consists of 10 cm line. One of the extremes presents a "no pain" indication and the other "unbearable pain". Each patient will be directed to mark with a single vertical dash the point that better matches his pain rating at the moment of the evaluation.

SECONDARY OUTCOMES:
Colour | In the first session and second session of the tooth whitening
  For a color rating before, immediately and 30 days after the bleaching treatment the spectrophotometer Vita Easy Shade will be used together with the Vita Classica scale, which will be organized from the highest value (B1) to the lowest (C4). To evaluate color with the spectrophotometer, first a mold will be made of the upper anterior teeth from canine to canine with heavy condensation silicone, which will serve as a guide to the spectrophotometer. A Window of 3 mm in diameter will be made on the vestibular face of the silicon guide in the area of the tooth where the color will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Reis, doctor, Principal Investigator — Universidade Estadual de Ponta Grossa
Locations (1):
- Universidade Estadual de Ponta Grossa, Guarapuava, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Charakorn P, Cabanilla LL, Wagner WC, Foong WC, Shaheen J, Pregitzer R, Schneider D. The effect of preoperative ibuprofen on tooth sensitivity caused by in-office bleaching. Oper Dent. 2009 Mar-Apr;34(2):131-5. doi: 10.2341/08-33. PMID 19363967
- [Derived] de Paula EA, Loguercio AD, Fernandes D, Kossatz S, Reis A. Perioperative use of an anti-inflammatory drug on tooth sensitivity caused by in-office bleaching: a randomized, triple-blind clinical trial. Clin Oral Investig. 2013 Dec;17(9):2091-7. doi: 10.1007/s00784-013-0918-2. Epub 2013 Jan 31. PMID 23371755